CLINICAL TRIAL: NCT00889083
Title: Evaluation of Hepatic Mitochondrial Function in Sepsis
Brief Title: Hepatic Mitochondrial Function in Sepsis
Status: Withdrawn | Type: Observational
Why Stopped: no patients to include
Sponsor: Professor C ICHAI (Other)
Responsible Party: Sponsor-Investigator, Professor C ICHAI, Professor Chair of IAAM, Institut d'Anesthesiologie des Alpes Maritimes
Organization: Institut d'Anesthesiologie des Alpes Maritimes (Other)
Other Study IDs: IAAM-2009-1
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Sepsis; Peritonitis
Keywords: Sepsis; Peritonitis; Mitochondria; Liver
MeSH Terms: conditions — Sepsis; Peritonitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Non septic patients needing hepatic surgery
- Sepsis: Septic patients needing surgery for peritonitis

SUMMARY:
Multi-organ failure due to sepsis is a major cause of death in critically ill patients. But the mechanisms leading to this condition are not fully understood. Mitochondrial dysfunction has been shown in skeletal muscle of critically ill septic patients. Liver is very important in sepsis as it is responsible of the synthesis of several inflammatory proteins. Moreover hepatic failure is associated to a bad outcome.

The aim of this study is to evaluate the hepatic mitochondrial function in sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Septic group : Peritonitis patients needing surgery
* Non septic group : Patients needing hepatic surgery

Exclusion Criteria:

* No liver biopsy performed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04 (Estimated); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Mitochondrial complex activities | during surgery

SECONDARY OUTCOMES:
Quantification of adenine nucleotides | during surgery
Quantification of oxidative stress markers | during surgery
Correlation between SOFA score and mitochondrial complex activities | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Carole Ichai, MD, PhD, Study Chair — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Background] Brealey D, Brand M, Hargreaves I, Heales S, Land J, Smolenski R, Davies NA, Cooper CE, Singer M. Association between mitochondrial dysfunction and severity and outcome of septic shock. Lancet. 2002 Jul 20;360(9328):219-23. doi: 10.1016/S0140-6736(02)09459-X. PMID 12133657
- [Background] Fredriksson K, Hammarqvist F, Strigard K, Hultenby K, Ljungqvist O, Wernerman J, Rooyackers O. Derangements in mitochondrial metabolism in intercostal and leg muscle of critically ill patients with sepsis-induced multiple organ failure. Am J Physiol Endocrinol Metab. 2006 Nov;291(5):E1044-50. doi: 10.1152/ajpendo.00218.2006. Epub 2006 Jun 27. PMID 16803854